CLINICAL TRIAL: NCT00884910
Title: Amendment on Phase 1 Trial N07VEG "Assessment of a Next Generation Indwelling Provox Voice Rehabilitation System (Vega)". Amendment 3: Long-term Use of the Provox Vega
Brief Title: Long Term Use of the Provox Vega 22.5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Atos Medical AB (Industry)
Collaborators: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: N07VEGA Amendment 22.5
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Results first posted 2010-11-03 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Total Laryngectomy
Keywords: laryngectomy; Provox Vega; voice prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Provox Vega voice prosthesis 22.5 Fr — The patients' current Provox2 voice prosthesis will be removed and the new Provox Vega voice prosthesis will be inserted.
  Other Names: indwelling voice prosthesis

SUMMARY:
The purpose of this study was to investigate the long-term feasibility of the new Provox Vega 22.5 voice prosthesis (outer diameter of 22.5 French) and its insertion system (SmartInserter) in laryngectomized patients who currently use a Provox2 voice prothesis.

DETAILED DESCRIPTION:
Nowadays, many laryngectomized patients use a voice prosthesis to speak. The Provox2 is an indwelling voice prosthesis that has been on the market since 1997. Recently a new Provox voice prosthesis has been developed, the Provox Vega. This prosthesis is available in 3 different outer diameters. In this study the device with an outer diameter of 22.5 French is tested. The Provox Vega 22.5 is the successor of the Provox2 voice prosthesis. Both prostheses have an outer diameter of 22.5 French.

Outcomes were recorded by means of patient questionnaires and device life.

It is expected that some patients will like the new device (Provox Vega 22.5) better than the old one (Provox2) because the airflow resistance for speaking of the new prosthesis is lower when measured in a laboratory.

ELIGIBILITY:
Inclusion Criteria:

* total laryngectomy
* Provox2 user
* at least two previous replacements

Exclusion Criteria:

* patients' refusal
* fistula problems
* Provox ActiValve users

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frans JM Hilgers, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited by the Netherlands Cancer Institute
Groups:
- Provox Vega 22.5: The newly developed Provox Vega voice prosthesis, with an outer diameter of 22.5 French, was placed in the tracheoesophageal puncture of laryngectomized patients. Before the study, the patients were using another voice prosthesis (Provox2). The Provox2 is the predecessor of the Provox Vega. At the start of the study the patients' Provox2 voice prosthesis was removed and replaced with the Provox Vega 22.5.
Period: Overall Study
Arm/Group | Provox Vega 22.5
Started | 33
Completed | 32 (patient diagnosed with primary pulmonary tumor during study)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Provox Vega 22.5
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 66.42 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 32
Region of Enrollment [Number; unit: patients]
  Netherlands | 33

OUTCOME MEASURES:

1. Secondary Outcome: Device Life Time
Description: Periodic replacement of voice prostheses is considered a normal event. Over time, the device is affected by Candida which may hinder closure of the valve flap. The device life time of the voice prosthesis is determined by leakage through the device that occurs because of incomplete closure of the valve flap. At the time of analysis (6 months after placement of the devices), 25 devices had been replaced because of leakage through the device and 8 devices were still in situ. The outcomes that are reported concern the 25 devices that had been replaced.
Time Frame: 6 months
Population: Six months after placement of the devices, 25 out of 33 had been replaced for leakage through the device. The median device life time is based on all 33 devices. The maximum of the range reflects the 6 months cut off and not the actual maximum device life time, because of the devices still in situ at the time of analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Provox Vega 22.5
Number analyzed (Participants) | 33
Days | 74 (60.8) [8 to 184]

2. Primary Outcome: Patient Preference
Description: Patients were asked "Which voice prosthesis do you prefer?" Answer options were "old one (Provox2)", "new one (Provox Vega 22.5)", or "no preference".
Time Frame: 3 months post insertion, or at end of device life (whichever comes sooner)
Population: All patients that participated in the study and finished it were analyzed
Measure: Number; unit: Patients
Arm/Group | Provox Vega 22.5
Number analyzed (Participants) | 32
Patients
  Provox Vega 22.5 | 14
  Provox2 | 7
  No preference | 11

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the entire period that the Provox Vega voice prosthesis was in place. Voice prostheses have a limited device life and need periodic replacement.
Description: Adverse events were assessed after the insertion procedure, upon notification of a problem by the patient, and when the Provox Vega needed replacement. Normal reasons for replacement (leakage through, size changes) were not considered adverse events.
Arm/Group | Provox Vega 22.5
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No